CLINICAL TRIAL: NCT03018717
Title: Randomized Multicenter Clinical Trial of a Integral Clinical Care Plan Shared With or Without Telemonitoring of Bio Constants in Patients With Chronic Diseases in Advanced Stages. ATLANTIC Project
Brief Title: Integral Clinical Plan Shared With or Without Telemonitoring of Constants in Patient With Chronic Diseases
Acronym: ATLAN_TIC01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Telefónica S.A. (Industry); Junta de Andalucia (Other Government); Salud Responde (Unknown)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATLAN_TIC01
Record Dates: First submitted 2016-12-12; First posted 2017-01-12 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2018-09

CONDITIONS: Chronic Lung Disease; Chronic Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tele-monitoring Constant (Other): To analyze the efficacy and cost-efficacy of incorporating tele-monitoring of bio-parameters into the shared comprehensive clinical care plan. Patients will receive in their home a kit consisting of a briefcase containing all equipment (scale, pulse-oximeter ... etc) and a logo access to devices (Tablet) through mobile communications m2m between patient and platform Management for Chronic Patients.
  Interventions: Other: Telemonitoring Constant
- Standard clinical care (Other): Standard clinical care plan shared between plan of attention to the patient with Pluri-pathological process and the care plan for patients with chronic diseases, based on a comprehensive clinical assistance shared between Primary Care and Hospital Care
  Interventions: Other: Standard clinical care

INTERVENTIONS:
Other: Telemonitoring Constant — telemedicine of Constant
  Arms: Tele-monitoring Constant
Other: Standard clinical care — The patient will self-monitor heart rate, blood pressure, weight, diuresis, and capillary glycemia (in the case of diabetes)
  Arms: Standard clinical care

SUMMARY:
Information and communications technologies (ICT) currently constitute a key element in the innovation and improvement of providing health-care to frail populations with advanced chronic diseases, but it´s efficacy, safety and cost-effectiveness has not yet been proven conclusively. The investigators are going to carry out a multi-center, randomized, parallel groups, phase III clinical trial in adult patient with heart and/or lung advanced diseases,aiming to analyze the efficacy and cost-efficacy of tele-monitorization of bio-parameters added to optimal standard of clinical care (shared clinical care plan) compared to the shared clinical care plan exclusively.

DETAILED DESCRIPTION:
a total number of 510 patients will be divided in 3 centers: Hospital University Virgen del Rocío; Hospital University Virgen Macarena and Public Hospital Comarcal of Serranía de Ronda. Patient will be randomized in Tele-monitoring Constant (TELEPAC) To analyze the efficacy and cost-efficacy of incorporating tele-monitoring of bio-parameters into the shared comprehensive clinical care plan or in Standard Clinical Care (PAC) based on a comprehensive clinical assistance shared between Primary Care and Hospital Care.

ELIGIBILITY:
Inclusion Criteria:

* Majority legal age (18 years of age or older)
* Present any of the following shortcomings:

Heart failure with baseline dyspnea ≥III of New York Heart Association (NYHA) Chronic respiratory insufficiency with basal dyspnea ≥III of Medical Research Council (MRC) Scale and / or oxygen saturation <90% and / or home oxygen therapy.

* Present Heart Failure or Respiratory Insufficiency with basal dyspnea grade <III (according to NYHA and MRC respectively) but have presented 2 or more income in the last year.
* Score of Patients with terminal or palliative medical diseases (score PALIAR) index between 0 and 7 points.
* To present one of the following assistance situations: hospital admission, follow-up in Home Hospitalization or Palliative Care Teams, specialized outpatient follow-up.
* Speak, understand, read and write Spanish, either the patient or the primary caregiver.
* Have basic knowledge of the use of mobile phones and applications of computer tablets (such knowledge will be confirmed by personal interview, with test of the device).
* Informed consent to participate in the study

Exclusion Criteria:

* Presence of malignant neoplastic disease ACTIVE except localized adenocarcinoma of prostate in hormonal treatment, and / or cutaneous basocellular-squamous cell carcinoma.
* In the case of Chronic Renal Disease if there is the possibility of entry into Substitutive Therapies (hemodialysis or transplantation)
* In the case of chronic liver disease, if there is a possibility of liver transplantation.
* Chronic neurological disease with established cognitive impairment (E. Pfeiffer with 7 or more errors and / or Mild cognitive evaluated (ECM with ≤18 points).
* Clinical situation of agony.
* Surprise question ("Would you be surprised if your patient died in the next 6 months?") With the result "I would not be surprised" + PALIAR Score Score ≥7.5 points.
* Participate in another tele-health initiative.
* Go simultaneously to a private health service and / or be institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2019-09-13 (Estimated)

PRIMARY OUTCOMES:
Reduce the number of hospital admissions and / or the number of hospital emergency visits and / or the number of primary care visits of the patients in the TELEPAC arm (patients with tele-monitoring) with respect to the PAC arm (patient without tele-Moni | Six month
  Monitoring number of hospitalizations and/or number of emergency visits in the period.

SECONDARY OUTCOMES:
Number of hospital admissions | six month
Safety by monitoring of adverse events and adverse clinical events related to the two arms of the clinical trial | six month
  analyze the safety of the two arms by monitoring the number of adverse events and adverse clinical events related to the two arms of the clinical trial.
quality of life related to health, of follow-up in both arms of the clinical trial, | At the time of inclusion, at 45 days and after 6 months of follow-up.
  Using a standardized Using a standardized questionnaire of quality of live related to health in adults (EQ-5D) adapted to Spanish.
quality of care and satisfaction perceived by the subjects in the two arms of the clinical trial. | at 45 days and after 6 months of follow-up
  Using the standardized questionnaire Service Performance (SERVPERF) adapted to health.
perceived quality and satisfaction with the technological instruments by the subjects in the two arms of the clinical trial. | at 45 days and after 6 months of follow-up,
  Using the Perceived quality for technical support (TSUQ) standardized questionnaire adapted
primary cost-effectiveness of the arm TELEPAC with respect to the arm PAC, using the incremental cost method. | six month
  using each of the patients that did not require hospital admission and / or emergency visits, as a unit of cost Of each patient.
To analyze the secondary incremental cost-effectiveness of the TELEPAC arm with respect to the PAC arm. | six month
  using each of the secondary efficacy variables as unit of cost and each patient's overall cost unit.
Number of admissions-visits to Hospital Emergency | six month
Number of visits to Primary Care Emergencies | six month
mortality | six month
Number of days of hospital stay | six month
Overall cost for patients in euros | six month

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Serranía de Ronda Hospital, Ronda, Málaga
  - Universitary Hospital Virgen Macarena, Seville, Seville
  - Universitary Hospital Virgen del Rocío, Seville, Seville
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario de Valme, Seville

IPD SHARING:
Plan to Share IPD: No